CLINICAL TRIAL: NCT04032054
Title: Comparison of Short Segment Mono-axial and Poly-axial Pedicle Screw Fixation for Thoracolumbar Fractures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Islam Mohamed Abd El Hameed, Resident doctor, Assiut University
Other Study IDs: TL pedicular screws fixation
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Spine Fracture
Keywords: thoracolumbar fractures
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- A: mono-axial
  Interventions: Device: mono-axial and poly-axial screws
- B: poly-axial
  Interventions: Device: mono-axial and poly-axial screws

INTERVENTIONS:
Device: mono-axial and poly-axial screws — types of pedicular screws for thoracolumbar fractures fixation

SUMMARY:
Comparison of short segment mono axial and poly axial pedicle screw fixation in thoracolumbar fractures regarding the best correction of the fracture and deformity and the maintenance of the correction.

DETAILED DESCRIPTION:
* Thoracolumbar spine trauma represents the most common area fractured in the spine In a large series of 3,142 patients with traumatic spinal fractures, Wang et al., 2012, reported that 54.9% of the patients had fractures in the thoracolumbar spine. Patients with complete neurological deficits generally have thoracic fractures, possibly due to a small canal diameter when compared to the cervical or lumbar spine Although grouped together, TLST is comprised of injures to the more rigid thoracic spine (T1-T10), the flexible and transitional thoracolumbar junction (T11-L2), more susceptible to injuries, and the lumbar spine L3-5. Early diagnosis and adequate management may improve patients' outcome and decrease its inherent disability.(1)
* Morphological classification of thoraco-lumbar fractures is based on the Magerl classification modified by the AOSpine Classification Group. For this evaluation radiograms and CT scans with multiplanar reconstructions are essential. In some cases additional MR images might be necessary.(2)
* The goal of fracture treatment is to obtain and maintain a stable reduction and early mobilization. A secondary aim is to restore sagittal alignment which has gained increasing emphasis in the last decade.(3)
* Posterior short segment fixation including the proximal and distal adjacent normal vertebrae is the most commonly performed surgery for the vast majority of thoracolumbar fractures, Posterior pedicle screw fixation has been shown to be simple, familiar, efficient, reliable, and safe for the reduction and stabilization of most fractures and remains the most popular technique.(4)
* The aim of our study is to compare between monoaxial short segment pedicle screw fixation and polyaxial short segment pedicle screw fixation

ELIGIBILITY:
Inclusion Criteria:

* Thoracolumbar fractures D4 - L3.
* Neurologically free.
* Age of the patients to be from 20 to 60 years.
* Type A3 and A4 according to the AO classification.

Exclusion Criteria:

* Pathological or Osteoporotic fractures.
* Lumbar degenerative diseases.
* Multisegement spine fractures.
* Poly traumatized patients

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: population will include all the recruited patients with thoracolumbar spine fracture eligible for our study according to inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
The sagittal cobb's angel. | base line
  the greatest angle at a particular region of the vertebral column, when measured from the superior endplate of a superior vertebra to the inferior endplate of an inferior vertebra.

SECONDARY OUTCOMES:
Vertebral body angel | base line
  the angel between upper and lower end plates of fractured vertebra
Anterior vertebral body height | base line
  distance between upper and lower end plates of same fractured vertebra